CLINICAL TRIAL: NCT01998074
Title: Evaluation of the Efficacy of a New Extensively Hydrolyzed Formula in Infants With Cow's Milk Protein Allergy
Brief Title: Evaluation of the Efficacy of a New Formula in Infants With Cow's Milk Protein Allergy
Acronym: Paradice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: UP2010-Paradice; BUN 143201010095 (Other: Commissie medische ethiek)
Record Dates: First submitted 2013-11-22; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Milk Hypersensitivity; Food Sensitivity; Protein Allergy
Keywords: Cow's Milk protein Allergy
MeSH Terms: conditions — Milk Hypersensitivity; Food Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study formula (Experimental)
  Interventions: Dietary Supplement: extensively hydrolyzed rice protein formula

INTERVENTIONS:
Dietary Supplement: extensively hydrolyzed rice protein formula

SUMMARY:
The aim of the study is to show the efficacy, tolerance and nutritional adequacy of a newly developed hydrolyzed rice formula in infants with a proven cow's milk protein allergy.

ELIGIBILITY:
Inclusion Criteria:

* Infants between 2 weeks and 6 months old
* In whom cow's Milk Protein Allergy has been proved by a food challenge performed during the previous month

Exclusion Criteria:

* Exclusively breast fed infants
* Preterm infants
* Infants already fed with an extensively hydrolyzed formula with no improvement of the symptoms.
* Infants fed an amino acid based formula
* Infants who had an anaphylactic reaction in the past

Ages: 2 Weeks to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Clinical improvement of symptoms of cow's milk protein allergy, through the use of a validated score | at 4 weeks

SECONDARY OUTCOMES:
Clinical improvement of symptoms of cow's milk protein allergy, through the use of a validated score | at 3 months
Clinical improvement of symptoms of cow's milk protein allergy, through the use of a validated score | at 6 months
Growth (weight, height, head circumference) | 1 month
Growth (weight, height, head circumference) | 3 months
Growth (weight, height, head circumference) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis, Brussels, Belgium

REFERENCES:
- [Derived] Vandenplas Y, De Greef E, Hauser B; Paradice Study Group; Paradice Study Group. An extensively hydrolysed rice protein-based formula in the management of infants with cow's milk protein allergy: preliminary results after 1 month. Arch Dis Child. 2014 Oct;99(10):933-6. doi: 10.1136/archdischild-2013-304727. Epub 2014 Jun 9. PMID 24914098